CLINICAL TRIAL: NCT02023983
Title: Official Title Verification of the Safety of Early Discharge (Within 72 Hours) in Low Risk Patients After Acute ST-segment Elevation Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention. Open Randomized Study.
Brief Title: Verification of the Safety of Early Discharge in Patients After Acute ST-segment Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamil Novobílský (Other)
Responsible Party: Sponsor-Investigator, Kamil Novobílský, M.D., Municipal Hospital Ostrava
Organization: Municipal Hospital Ostrava (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KN-11-2013
Record Dates: First submitted 2013-12-16; First posted 2013-12-30 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction With ST-segment Elevation; Primary Percutaneous Coronary Intervention; Early Discharge
Keywords: ST-segment elevation myocardial infarction; Primary percutaneous coronary intervention; Low risk; Early discharge
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early discharge (Experimental)
  Interventions: Other: Early discharge
- Standard discharge (Active Comparator)
  Interventions: Other: Standard discharge

INTERVENTIONS:
Other: Early discharge — Early discharge (within 72 hours) of selected patients with low risk of complications after myocardial infarction with ST segment elevation, treated with successful percutaneous coronary intervention
  Arms: Early discharge
Other: Standard discharge — Discharge after myocardial infarction with ST segment elevation in a standard way accordingly with present practice and physician´s decision (usually 4th-7th day)
  Arms: Standard discharge

SUMMARY:
The aim of the study is to prove that early discharge (within 72 hours) in selected group of patients after myocardial infarction with elevations of ST-segment is feasible and safe

DETAILED DESCRIPTION:
The aim of the study is to prove

* that early discharge (within 72 hours) in selected group of patients with low risk of follow-up complications after myocardial infarction with elevations of ST-segment, treated with primary percutaneous coronary intervention, is feasible and safe
* that early discharge is comparable with the group of patients, discharged in a standard way accordingly with present practice and physician´s decision (usually 4th-7th day), thus it is not associated with higher incidence of complications in 90th day after myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 do ≤ 75 years
* Acute myocardial infarction with ST-segment elevation, treated with successful percutaneous coronary intervention within 12 hours from the onset of symptoms
* Left ventricle ejection fraction ≥ 45% by echocardiography
* Single- or two-vessel disease (stenosis of major epicardial artery ≥ 70%)
* Haemodynamic and rhythmic stability (Killip class I, no arrythmia requiring treatment occurring > 2 hours after PCI)
* Assumed good cooperation and social background

Exclusion Criteria:

* Symptoms of residual ischemia
* Significant comorbidities or abnormalities in paraclinical tests, requiring additional evaluation within continuing hospitalization
* Contraindication of dual antiplatelet therapy or need for anticoagulation therapy
* Hihg risk of bleeding complications
* Participation in other clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal Hospital Ostrava, Ostrava, Czechia

REFERENCES:
- [Derived] Novobilsky K, Stipal R, Cerny P, Horak I, Kaucak V, Mrozek J, Vaclavik J, Kryza R. Safety of early discharge in low risk patients after acute ST-segment elevation myocardial infarction, treated with primary percutaneous coronary intervention. Open label, randomized trial. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2019 Feb;163(1):61-66. doi: 10.5507/bp.2018.041. Epub 2018 Aug 28. PMID 30181666

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Discharge | Standard Discharge
Started | 76 | 75
Completed | 76 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Discharge | Standard Discharge | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 18 | 19 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 61 | 63 | 124
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 41 | 41 | 82
Diabetes [Count of Participants; unit: Participants] | 7 | 7 | 14
Impaired glucose tolerance [Count of Participants; unit: Participants] | 8 | 12 | 20
Hyperliporoteinemia [Count of Participants; unit: Participants] | 54 | 58 | 112
Previous myocardial infarction [Count of Participants; unit: Participants] | 3 | 6 | 9
Previous PCI [Count of Participants; unit: Participants] | 2 | 6 | 8
Previous stroke / transient ischemic attack [Count of Participants; unit: Participants] | 2 | 2 | 4
Peripheral arterial disease [Count of Participants; unit: Participants] | 2 | 1 | 3
Smoking [Count of Participants; unit: Participants] | 56 | 45 | 101
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (5.1) | 27.3 (3.5) | 28.64 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Composite of Incidence of Death, Reinfarction, Unstable Angina Pectoris, Stroke, Unplanned Rehospitalization, Repeat Target Vessel Revascularization and Stent Thrombosis in 90 Days After Myocardial Infarction (MI)
Description: Fischer´s exact test was used for comparison of qualitative variables between two groups. For comparison of quantitative variables we applied Mann-Whitney U test, respectively Student´s t-test (age). Normality of data was assessed with Shapiro-Wilk test. Values of p < 0.05 were considered as statistically significant.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Early Discharge | Standard Discharge
Number analyzed (Participants) | 76 | 75
Participants
  Primary composite endpoint | 5 | 6
  Death | 0 | 0
  Myocardial infarction | 1 | 2
  Unstable angina | 1 | 1
  Unplanned rehospitalization | 5 | 6
  Repeated target vessel revascularization | 1 | 3
  Stent thrombosis | 0 | 2
  Stroke | 0 | 0
Statistical Analysis 1: Comparison: Early Discharge vs Standard Discharge; Test type: Other; p = 0.765, Fisher Exact

2. Secondary Outcome: Complications Associated With the Puncture Site Requiring Treatment in 30 Days After Myocardial Infarction (MI)
Description: as for outcome 1
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Early Discharge | Standard Discharge
Number analyzed (Participants) | 76 | 75
Participants | 1 | 0
Statistical Analysis 1: Comparison: Early Discharge vs Standard Discharge; Test type: Other; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: 90 days
Description: Definitions of adverse event and serious adverse event meet the clinicaltrials.gov Definitions
Arm/Group | Early Discharge | Standard Discharge
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 5/76 | 6/75
Other Adverse Events (participants affected / at risk) | 1/76 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Discharge (N=76) | Standard Discharge (N=75)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Unstable angina (Cardiac disorders) | 1 (1) | 1 (1)
Brain cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Discharge (N=76) | Standard Discharge (N=75)
Radial artery occlusion (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitation of the study is limited number of probands enrolled in one centre.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-08-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT02023983/Prot_SAP_001.pdf
  • Informed Consent Form (2013-08-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT02023983/ICF_002.pdf